CLINICAL TRIAL: NCT01829152
Title: Verizon Wireless - Sarasota Memorial Hospital Converged Health Management (CHM) For Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Verizon Wireless (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: SARHF-0319
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Heart Failure
Keywords: heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Subjects in the Control Group will receive Heart Failure care as routinely delivered by the SMH HF clinicians according to their standards of care.
- CHM Intervention Group (Experimental): The Intervention Group subjects will receive Converged Health Management (CHM) in addition to continuing to receive care as routinely delivered by the SMH HF clinicians.
  Interventions: Device: CHM

INTERVENTIONS:
Device: CHM
  Arms: CHM Intervention Group

SUMMARY:
The primary objective is to evaluate the impact on heart failure related quality of life when integrating a mobile health system, Verizon Wireless's Converged Health Management (CHM), into a subject's self-management of their heart failure (HF) as well as in the medical management of HF by the subjects' clinical team.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥ 18 years of age)
2. A least 1 prior hospitalization within the past 12 months for HF based upon the presence of at least 1 symptom (dyspnea, orthopnea, or edema) AND at least 1 sign (rales, peripheral edema, ascites, or pulmonary vascular congestion on chest radiography)AND treatment with a loop diuretic during the hospital stay OR Symptoms of New York Hospital Association (NYHA) Class 2+ symptoms: dyspnea, fatigue, or chest pain with normal physical activity (class II), less than ordinary activity (class III) or at rest (class IV).

   Information may be provided by subject self-report obtained during the initial screening process and/or by medical record confirmation. Compliance with all eligibility criteria will be confirmed at the initial study visit before subject is presented with the ICF.
3. Receiving care at the SMH HF Clinic and assessed by the clinic at least twice. (Those who were seen in person on their first visit and then followed-up by telephone thereafter will be considered eligible).
4. Able to provide contact information for someone who agrees to provide information about the subject if the subject is not available to do so.
5. Capability of understanding and willingness to comply with the protocol and study requirements, assessed according to the Principal Investigator's judgment.
6. Ability to understand and willingness to sign a written informed consent document, assessed according to the Principal Investigator's judgment.

Exclusion Criteria:

1. Decline to participate in the study
2. Reside in an area with limited to no Verizon Wireless coverage as determined by VZ using the VZ zip code coverage analysis technology.
3. Scheduled procedure for left ventricular device implantation, or listed for potential cardiac transplant
4. Current resident of a long-term care or skilled nursing facility
5. Currently receiving palliative or hospice care
6. Human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS) based on past medical history or subject self-report
7. Dialysis-dependent, end-stage renal disease
8. A concurrent physical condition (including rare or chronic diseases such as sickle cell anemia or cystic fibrosis) or mental health condition (including dementia, schizophrenia, or other mental illness) that in the view of the Principal Investigator would compromise the subject's ability to fulfill the protocol requirements or affect the subject's safety during the study
9. Are unable or unwilling to comply with the study requirements as instructed including coming to the SMH HF clinic for the 2 study visits.
10. For subjects in the Intervention Group that are:

    1. Unable or unwilling to return to the SMH clinic to receive their training, devices and study material after signing the informed consent form and being randomized into the Intervention Group;
    2. Unable or unwilling to use the biometric devices and CHM at least one time per day.
11. Are pregnant or planning to become pregnant during the study.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Quality of life, as measured by subject response to the Minnesota Living with Heart Failure Questionnaire (MLWHF). | 6 months

SECONDARY OUTCOMES:
To assess the impact of the CHM intervention on the subjects' medication adherence as gathered from the Morisky Medication Adherence questionnaire. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Voelker, MD, Principal Investigator — Sarasota Memorial Hospital
Locations (1):
- Sarasota Memorial Hospital Heart Failure Clinic, Sarasota, Florida, United States